CLINICAL TRIAL: NCT06400160
Title: An Open-label, Multi-center, and Dose-escalation, Phase 1/2a Clinical Trial to Assess the Maximum Tolerated Dose(MTD), Safety, and the Anti-tumor Effect of TB511 Monotherapy in Patients With Advanced Solid Tumors Refractory or Intolerant to Standard of Care(SoC) and Pembrolizumab Combination Therapy in Patients With Advanced Solid Tumors Relapsed or Refractory
Brief Title: Clinical Trial of TB511 in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Twinpig Biolab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB001 Version 2.1_2024-10-25
Record Dates: First submitted 2024-04-01; First posted 2024-05-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; Prostate Cancer; Colorectal Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: An Open-label, Multi-center, and Dose-escalation, Phase I/IIa Clinical Trial to Assess the Maximum Tolerated Dose (MTD), Safety, and the Anti-tumor Effect of TB511 Monotherapy in Patients with Advanced Solid Tumors Refractory or Intolerant to Standard of Care (SoC) and Pembrolizumab Combination Therapy in Patients with Advanced Solid Tumors Relapsed or Refractory
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TB511 (Experimental): * Product name or code: TB511 Injection (8 mg)
    * Formulation and appearance: White or off-white color of lyophilized powder ③ Main ingredient: TB511 ④ Storage method: Store in a hermetic container in a freezer (-20℃); protect from light
  Interventions: Drug: TB511
- Concomitant drug (Other): * Product name or code: Keytruda
    ② Formulation and appearance: An injection comprised of clear to slightly opalescent, colorless to slightly yellow liquid contained in a colorless and transparent vial.
    ③ Main ingredient: Pembrolizumab
  * Storage method: Store in a hermetic container, refrigerated at 2 to 8℃; protect from light; do not freeze
  Interventions: Drug: Keytruda

INTERVENTIONS:
Drug: TB511 — TB511 is a peptide drug conjugate (PDC) which composed of TAMpep826 peptide. TB511 is a white amorphous powder used for subcutaneous injections. TB511 is a peptide drug conjugate that combines a transporter peptide with a specific targeting of M2 macrophages and an apoptosis-inducing peptide (dKLA). As a transporter, the M2 binding peptide acts as a drug conjugate, explicitly binding to M2 macrophages and inducing cell penetration. In the cells, the dKLA component of TB511 binds to the mitochondrial membrane, destroys the mitochondrial membrane, and induces apoptosis by causing cytochrome release, leading to the destruction of the mitochondria and subsequent death of M2 macrophages.
  Arms: TB511
Drug: Keytruda — KEYTRUDA binds to the PD - 1 receptor, blocking both immune-suppressing ligands, PD L1 and PD L2, from interacting with PD - 1 to help restore T-cell response and immune response.
  Arms: Concomitant drug

SUMMARY:
1. Study population

   [TB511 Monotherapy Cohort for Phase 1 and Phase 2a Clinical Trial] Patients with advanced solid tumors who are either refractory or intolerant to standard of care (SoC).

   [Immune checkpoint inhibitors (ICIs) Combination Therapy Cohort for Phase 2a Clinical Trial] Patients with advanced solid tumors who are refractory to immune checkpoint inhibitors (ICIs) such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 inhibitors or who have no available standard of care.
2. Objectives of the Clinical Trial

2.1 Primary Objectives [Phase 1 Clinical Trial]

* To evaluate the safety and tolerability of TB511 monotherapy in patients with advanced solid tumors and to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D).

[Phase 2a Clinical Trial]

* To evaluate the Objective Response Rate (ORR) of TB511 monotherapy and TB511 in combination with Pembrolizumab in patients with advanced solid tumors (based on Response Evaluation Criteria In Solid Tumors Version 1.1, RECIST v1.1).

2.2 Secondary Objectives [Phase 1 Clinical Trial]

* To evaluate the safety of TB511 monotherapy.
* To assess the Objective Response Rate (ORR) and anti-tumor activity of TB511 monotherapy (based on RECIST v1.1).
* To characterize the pharmacokinetic (PK) profile of TB511 monotherapy.

[Phase 2a Clinical Trial]

* To evaluate the Disease Control Rate (DCR), Duration of Response (DoR), and Progression-Free Survival (PFS) of TB511 monotherapy and TB511 in combination with Pembrolizumab.
* To assess the safety and tolerability of TB511 monotherapy and TB511 in combination with Pembrolizumab.
* To characterize the pharmacokinetic (PK) profile of TB511 monotherapy and TB511 in combination with Pembrolizumab.

2.3 Exploratory Objectives

* To compare changes in biomarker levels of TB511 monotherapy.
* To assess immunogenicity of TB511 by measuring anti-drug antibodies (ADA).

DETAILED DESCRIPTION:
1. Number of participants

   [Phase 1 Clinical Trial] 3 to 6 patients per dose group

   [Phase 2a Clinical Trial] Approximately 20 patients per cohort (Cohort 1: Approximately 20 patients, Cohort 2: Approximately 20 patients)
2. Study Duration

   * Total clinical trial duration: Approximately 36 months from the date of IRB approval (however, this may be adjusted depending on the enrollment rate of participants.)
   * Participation duration for individual participants
   * Screening period: Up to 4 weeks (28 days)
   * Treatment period: Each cycle consists of 3 weeks (21 days), and administration will continue until a reason for discontinuation occurs.
   * Safety follow-up period: 6 weeks after the End of Treatment (EOT)
3. Investigational Product

<!-- -->

1. Study drug

   * Product name or code: TB511 Injection (8 mg)

     * Formulation and appearance: White or off-white color of lyophilized powder ③ Main ingredient: TB511 ④ Storage method: Store in a hermetic container in a freezer (-20℃); protect from light
2. Concomitant drug

   * Product name or code: Keytruda

     * Formulation and appearance: An injection comprised of clear to slightly opalescent, colorless to slightly yellow solution contained in a colorless and transparent vial.

       * Main ingredient: Pembrolizumab ④ Storage method: Store in a hermetic container, refrigerated at 2 to 8℃; protect from light; do not freeze

         4. Dosage and method of administration

[Phase 1 Clinical Trial]

1. TB511

   * Starting Dose group: 4 mg

     * Dose Escalation groups: 4 mg, 8 mg, 16 mg, 24 mg

       ③ Dose De-escalation: 12 mg, 20 mg

       ④ Administration method: 1 cycle consists of 3 weeks (21 days). TB511 will be administered subcutaneously into the abdomen once every 7 days for 3 weeks (21 days). Repetitive injections at the same site should be avoided; instead, rotate injection sites within the abdominal area. Do not inject into sensitive or abnormal skin areas (e.g., wounds, rashes, redness, induration, etc.).

       ⑤ Administration Plan: Administration will continue until unacceptable toxicity, disease progression (PD) per RECIST v1.1, or other reasons requiring discontinuation occur.

[Phase 2a Clinical Trial]

1. TB511

   * Dose: Recommended dose for Phase 2a determined in Phase 1.

     ② Administration method: 1 cycle consists of 3 weeks (21 days). TB511 will be administered subcutaneously into the abdomen once every 7 days for 3 weeks (21 days). Repetitive injections at the same site should be avoided; instead, rotate injection sites within the abdominal area. Do not inject into sensitive or abnormal skin areas (e.g., wounds, rashes, redness, induration, etc.).

     ③ Administration Plan: Administration will continue until unacceptable toxicity, disease progression (PD) per RECIST v1.1, or other reasons requiring discontinuation occur.
2. Pembrolizumab

   * Dose: 200 mg or dose adjusted according to the approved labeling.

     ② Administration Method: Pembrolizumab is administered by continuous intravenous infusion for 30 minutes, once every 3 weeks (When used in combination with TB511, Pembrolizumab should be administered first, followed by TB511 at least 30 minutes later).
     * Administration Plan: Administration will continue until unacceptable toxicity, disease progression (PD) per RECIST v1.1, or other reasons requiring discontinuation occur.

       5. Study Method

This clinical trial consists of a Phase 1 dose-escalation study to determine the maximum tolerated dose (MTD) of TB511 and establish the recommended Phase 2a dose (RP2D) in patients with advanced solid tumors who are refractory or intolerant to standard of care, and a Phase 2a study to evaluate the anti-tumor effect of TB511 monotherapy in dose determined in Phase 1 (Cohort 1) and TB511 in combination with Pembrolizumab (Cohort 2) in patients with advanced solid tumors for whom no standard of care is available, including those who are refractory to immune checkpoint inhibitors (ICIs) such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 agents or who have experienced disease progression.

Participants who voluntarily sign the written informed consent form will undergo screening tests to assess eligibility during the screening period. Subjects who meet all inclusion and none of the exclusion criteria will be enrolled in this clinical trial and receive the investigational product at the assigned dose level. 1 cycle of administration of the investigational product is 3 weeks (21 days), and enrolled participants continue to receive the investigational product until intolerable toxicity, verification of progressive disease (PD) as defined by RECIST v1.1, or any other reason for discontinuing administration occur. Tumor response assessments (CT/MRI) will be conducted on Day 1 of Cycle 1 and every 2 cycles thereafter. Pharmacokinetic (PK) evaluation will be performed on Day 1 and Day 15 of Cycle 1, and exploratory evaluation will be performed during screening, and on Day 8 and Day 15 of Cycle 1.

[Phase 1 Clinical Trial - TB511 Monotherapy] The Phase I clinical trial will follow a 3+3 design, starting from the lowest dose cohort and continuing until the maximum tolerated dose (MTD) is determined. Depending on the MTD determination method, 3 to 6 participants will be sequentially enrolled in each dose-escalation level (TB511: 4 mg, 8 mg, 16 mg, 24 mg) with at least a 3-day interval and TB511 is administered for 1 cycle to determine dose limiting toxicity(DLT). DLT assessment will be conducted in Cycle 1. Dose escalation or de-escalation will be decided by the Safety Review Committee (SRC) after the completion of DLT evaluation of the last participant in each dose level. If no DLT is observed, the study will proceed to the next higher dose level. If DLT occurs, the trial may proceed with an intermediate dose level, as defined below. After completion of dose escalation or de-escalation, the Recommended Phase 2a Dose (RP2D) will be determined based on the MTD and overall toxicity evaluation. The SRC will also decide whether to continue or discontinue the trial.

<Dose De-escalation Scheme>

If DLT is observed at a given dose level, the dose will be de-escalated to an intermediate dose* as follows:

- If toxicity occurs at 24 mg, the intermediate dose will be 20 mg.

* If toxicity occurs at 16 mg, the intermediate dose will be 12 mg.

  * Intermediate dose: An intermediate dose between the given dose level and one-step lower dose level.

ELIGIBILITY:
Inclusion Criteria:

[Common]

1. Male and female adults who are 19 years old or older at the time of obtaining informed consent form.
2. Patients with at least one measurable lesion by RECIST v1.1.
3. Patients whose Eastern Cooperative Oncology Group Performance Status (ECOG PS) is 0 or 1.
4. Female patients of childbearing potential who have not undergone sterilization surgery must agree to use appropriate contraception* for 6 months after the end of administration of the investigational product and must satisfy one of the following conditions at the time of screening to establish that they are not pregnant.

   • Women over the age of 50 who have had amenorrhea for at least 12 months after the termination of all exogenous hormone treatment.
   * Documented irreversible surgical sterilization by hysterectomy, dual ovariectomy, or oophorectomy (tubal litigation does not satisfy this criteria)
   * Women under the age of 50 who have had amenorrhea for at least 12 months after the termination of all exogenous hormone treatment and whose luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the post-menopause range determined by the clinical trial institution.
5. Male patients who have not undergone vasectomy must agree to use a barrier method of contraception (i.e., condom) and agree that both they and their partners will use an appropriate method of contraception* through 6 months after the end of administration of the investigational product.

   *Appropriate methods of contraception include: complete abstinence, hormonal contraceptives not known to have drug interactions [levonorgestrel-releasing intrauterine system (IUS) (e.g., Mirena), medroxyprogesterone (e.g., Provera)], copper intrauterine device, and partner's vasectomy. Periodic abstinence (e.g., calendar-based, ovulation tracking, or basal body temperature methods) and withdrawal are not considered appropriate methods of contraception.
6. Patients who have been provided with sufficient explanations on this clinical trial, have voluntarily decided to participate in this clinical trial and have agreed in writing to faithfully comply with the requirements of the clinical trial.

[Cohort of TB511 Monotherapy in Phase 1 and Phase 2a Clinical Trials]

1) Patients with cytologically or histologically confirmed advanced solid tumors who are either refractory or intolerant to standard of care (SoC).

[Cohort of ICIs Combination Therapy in Phase 2a Clinical Trial] 1) Patients with advanced solid tumors who, at the time of screening, are refractory to or have experienced disease progression during treatment with immune checkpoint inhibitors (ICIs) such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 agents within their approved indications, and for whom no standard therapy is available.

- This includes: melanoma, non-small cell lung cancer, head and neck cancer, classical Hodgkin lymphoma, urothelial carcinoma, gastric cancer, esophageal cancer, renal cell carcinoma, endometrial cancer, microsatellite instability-high (MSI-H) cancer, MSI-H colorectal cancer, triple-negative breast cancer, cervical cancer, biliary tract cancer, and hepatocellular carcinoma.

Exclusion Criteria:

[Common] Current Disease and Medical History

1. Patients who have had other malignant tumors within 5 years prior to the screening (provided, however, that patients with basal cell carcinoma that requires only stable long-term follow-up without treatment can be enrolled).
2. Patients who had been subject to chemotherapy, radiotherapy, or biological therapy within 4 weeks prior to the screening.
3. Patients who had undergone major surgery requiring general anesthesia within 4 weeks prior to the screening.
4. Patients with brain metastasis who have symptoms or required treatment (provided, however, that patients with asymptomatic metastasis that does not require treatment [excluding anticonvulsants used in maintenance therapy] can be enrolled).
5. Patients with systemic disease for which administration of anti-cancer drugs is deemed inappropriate by the investigator.
6. Patients with the following cardiovascular disease at the screening

   * Myocardial infarction, unstable angina, stroke, or transient ischemic within 6 months.
   * QTc interval ≥ 480 msec or clinically significant electrocardiographic change.
   * Congestive heart failure classified as New York Heart Association (NYHA) class III or above.
7. Patients who are HIV-positive.
8. Patients whose participation in the clinical trial is deemed inappropriate by the investigator based on their results of Hepatitis B virus and Hepatitis C virus test.(Not applicable to patients with hepatocellular carcinoma.)

   However, the following cases are allowed:
   * For patients positive for HBsAg or HBcAb: HBV DNA must be ≤ 2000 IU/mL or undetectable.
   * For patients positive for HCV Ab: HCV RNA must be negative or the patient must have completed antiviral treatment and be stabilized.
9. Patients with acute or severe hepatitis.
10. Patients with autoimmune disease or with history of chronic or recurrent autoimmune disease.
11. Patients with history of organ transplantation.
12. Patients with history of identical hematopoietic stem cell transplantation.
13. Patients with history of interstitial pneumonia requiring steroid treatment.
14. Patients with known hypersensitivity to recombinant drugs (drugs with active ingredients of peptide or protein).
15. Patients with history of hypersensitivity to the components of TB511.

    Prohibited Drugs
16. Patients who require continuous treatment with immunosuppressants or systemic corticosteroid administration (Note: Use of topical corticosteroids such as intra-articular, intranasal, ophthalmic, or inhaled formulations is permitted. Temporary use of systemic corticosteroids administration for the treatment or prevention of contrast agent allergies or adverse reactions is also allowed.)
17. Patients who have received live or attenuated live vaccines within 4 weeks prior to the screening.

    Laboratory tests
18. Patients with the following laboratory levels at the time of screening.

    * ANC < 1,500/mm³
    * Platelet count < 100,000/mm³ (for hepatocellular carcinoma: < 75,000/mm³)
    * Hemoglobin < 9.0 g/dL (Patients can be enrolled if hemoglobin level is recovered to ≥ 9.0 g/dL during the screening period; however, blood transfusion within 7 days prior to the screening to fulfill this criterion is not allowed.)
    * AST, ALT > 3 × ULN (provided, however, that if liver metastasis is involved, AST, ALT > 5 × ULN)
    * Total bilirubin > 1.5 × ULN
    * Serum creatinine > 1.5 × ULN

    Others
19. Pregnant, breastfeeding women, or patients with a positive pregnancy test at the time of screening.
20. Patients who, in the investigator's judgment, have an expected survival of less than 12 weeks.
21. Patients who have received other investigational drugs within 4 weeks prior to screening (Patients who did not receive investigational products or who participated only in non-interventional observational studies can be eligible).
22. Any patient deemed unsuitable for participation in this clinical trial at the discretion of the investigator.

[Only applicable to the cohort of TB511 and ICIs combination therapy in Phase 2a Clinical Trial]

1. Patients with thyroid-stimulating hormone (TSH) levels above the institutional upper limit of normal (ULN) at the time of screening (Note: patients with abnormal TSH levels may be eligible if free T4 and total T3 levels are within normal ranges).
2. Patients with a history of hypersensitivity to any component of pembrolizumab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase I Clinical trial-Maximum tolerated dose (MTD). | 1 year
  1. Definition and Assessment of Dose Limiting Toxicity (DLT) DLT is an adverse event or abnormal laboratory level unrelated to the progress of the disease or intercurrent disease that limits dose escalation and is consistent with one or more of the following criteria: DLT assessment is conducted only at Cycle 1 after completion of Cycle 1. However, even during Cycle 1, DLT can be immediately evaluated if toxicity is determined to be DLT. DLT assessment is conducted in accordance with NCI-CTCAE v5.0 based on individual assessment items on hematological/non-hematological toxicity and other toxicities.
  2. Definition and Determination of Maximum Tolerated Dose (MTD) When 2 out of 3 subjects or 2 out of 6 subjects experience DLTs, the dose is considered intolerable, the subsequent dose escalation is stopped, and a level lower than the dose is declared the maximum tolerable dose (MTD).
Phase I Clinical trial-Recommended Phase IIa dose (RP2D). | 1 year
  RP2D of Phase IIa clinical trial is determined through MTD and overall toxicity assessment.
Phase IIa Clinical trial-anti-tumor effect-to evaluate the Objective response rate (ORR) of TB511 monotherapy and combination therapy with Pembrolizumab in patients with advanced solid tumors (based on RECIST v1.1). | 2 years
  Solid tumor response is evaluated in accordance with RECIST v1.1 and immune RECIST (iRECIST).
  Objective response rate (ORR): Fraction of subjects whose best overall response is Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Phase I clinical trial-anti-tumor effects of TB511 Monotherapy-the Objective response rate (ORR) | 1 year
  Solid tumor response is evaluated in accordance with RECIST v1.1. Objective response rate (ORR): Fraction of subjects whose best overall response is Complete Response (CR) or Partial Response (PR)
Phase I clinical trial-anti-tumor effects of TB511 Monotherapy-Disease control rate (DCR) | 1 year
  Disease control rate (DCR): Fraction of subjects whose best overall response is CR, PR or Stable Disease (SD)
Phase I clinical trial-anti-tumor effects of TB511 Monotherapy-Duration of response (DoR) | 1 year
  Duration of response (DoR): From the point of time when response occurs to (CR or PR) PD or death due to any reason.
Phase I clinical trial-safety-adverse events of TB511 Monotherapy | 1 year
  Safety Assessment and Method of Assessment
  1) Adverse Events Adverse events are a general term for symptoms, signs, and abnormal values of laboratory tests that occur or worsen after the administration of an investigational product. The AE name, onset/end dates, severity, treatment and outcomes, and relationship to the investigational product should be documented in the AE pages of the eCRFs.
Phase I clinical trial-safety-vital signs of TB511 Monotherapy | 1 year
  2) Vital signs Findings of vital signs that meet the definitions of AEs after the administration of the investigational product should be reported as AEs.
Phase I clinical trial-safety-physical examination and ECG of TB511 Monotherapy | 1 year
  3) Physical examination and ECG After the administration of the investigational product, findings in physical examinations that meet the definitions of AEs or ECGs showing clinically significant changes should be reported as AEs.
Phase I clinical trial-safety-laboatory test of TB511 Monotherapy | 1 year
  4) Laboratory test Laboratory test results will be categorized into normal or abnormal (NCS or CS). Any result after the administration of the investigational product showing clinically significant changes from baseline should be reported as AEs.
PK parameters for TB511 (Area Under the Curve from 0 to 24 h (AUC)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 AUC
PK parameters for TB511 (AUC to the Last Measurable Concentration from 0 to 24 h (AUClast)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 AUClast
PK parameters for TB511 (Area under the plasma concentration-time curve extrapolated to infinity from 0 to 24 h (AUCinf)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 AUCinf
PK parameters for TB511 (Peak Plasma Concentration from 0 to 24 h (Cmax)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 Cmax
PK parameters for TB511 (Time to Obtain Maximum Plasma Concentration from 0 to 24 h (Tmax)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 Tmax
PK parameters for TB511 from 0 to 24 h (half-life (t1/2)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 half-life (t1/2)
PK parameters for TB511 (Clearance from 0 to 24 h (CL/F)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 CL/F
PK parameters for TB511 (Volume of distribution from 0 to 24 h (Vd/F)) [Time Frame: Day 1 of first 1 cycle] | 1 year
  Determine TB511 Vd/F
PK parameters for TB511 (Area Under the Curve from 0 to 24 h at steady-state (AUCss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 AUCss
PK parameters for TB511 (AUC to the Last Measurable Concentration from 0 to 24 h at steady-state (AUClast ss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 AUClast, ss
PK parameters for TB511 (Area under the plasma concentration-time curve extrapolated to infinity from 0 to 24 h at steady-state (AUCinf, ss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 AUCinf, ss
PK parameters for TB511 (Peak Plasma Concentration from 0 to 24 h at steady-state (Cmax ss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 Cmax, ss
PK parameters for TB511 (Time to Obtain Maximum Plasma Concentration from 0 to 24 h at steady-state (Tmax, ss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 Tmax, ss
PK parameters for TB511 (half-life from 0 to 24 h at steady-state (t1/2, ss)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 half-life (t1/2, ss)
PK parameters for TB511 (Clearance from 0 to 24 h at steady-state (CL, ss/F)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 CL, ss/F
PK parameters for TB511 (Volume of distribution from 0 to 24 h at steady-state (Vd, ss/F)) [Time Frame: Day 21 of first 1 cycle] | 1 year
  Determine TB511 Vd, ss/F
Phase IIa-anti-tumor effects of TB511 Monotherapy and TB511 & pembronizumab compination therapy-Disease control rate (DCR) | 2 years
  Disease control rate (DCR): Fraction of subjects whose best overall response is CR, PR or SD
Phase IIa-anti-tumor effects of TB511 Monotherapy and TB511 & pembronizumab compination therapy-Duration of response (DoR) | 2 years
  Duration of response (DoR): From the point of time when response occurs to (CR or PR) PD or death due to any reason.
Phase IIa-anti-tumor effects of TB511 Monotherapy and TB511 & pembronizumab compination therapy-Progression-free survival (PFS) period | 2 years
  Progression-free survival (PFS) period: Period from the initial date of administration of the investigational product to the date when objective progressive disease (PD) is verified by the investigator, or the date of death, whichever occurs first.
Phase IIa-the safety-adverse events of TB511 Monotherapy and TB511 & pembronizumab compination therapy | 2 years
  1) Adverse Events Adverse events are a general term for symptoms, signs, and abnormal values of laboratory tests that occur or worsen after the administration of an investigational product. The AE name, onset/end dates, severity, treatment and outcomes, and relationship to the investigational product should be documented in the AE pages of the eCRFs.
Phase IIa-the safety-vital signs of TB511 Monotherapy and TB511 & pembronizumab compination therapy | 2 years
  2) Vital signs Findings of vital signs that meet the definitions of AEs after the administration of the investigational product should be reported as AEs.
Phase IIa-the safety-Physical examination and ECG of TB511 Monotherapy and TB511 & pembronizumab compination therapy | 2 years
  3) Physical examination and ECG After the administration of the investigational product, findings in physical examinations that meet the definitions of AEs or ECGs showing clinically significant changes should be reported as AEs.
  Findings of vital signs that meet the definitions of AEs after the administration of the investigational product should be reported as AEs.
Phase IIa-the safety-Laboratory test of TB511 Monotherapy and TB511 & pembronizumab compination therapy | 2 years
  4) Laboratory test Laboratory test results will be categorized into normal or abnormal (NCS or CS). Any result after the administration of the investigational product showing clinically significant changes from baseline should be reported as AEs.
PK parameters for TB511 and Pembrolizumab combination (Area Under the Curve from 0 to 24 h (AUC)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUC
PK parameters for TB511 and Pembrolizumab combination (AUC to the Last Measurable Concentration from 0 to 24 h (AUClast)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUClast
PK parameters for TB511 and Pembrolizumab combination (Area under the plasma concentration-time curve extrapolated to infinity from 0 to 24 h (AUCinf)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUCinf
PK parameters for TB511 and Pembrolizumab combination (Peak Plasma Concentration from 0 to 24 h (Cmax)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Cmax
PK parameters for TB511 and Pembrolizumab combination (Time to Obtain Maximum Plasma Concentration from 0 to 24 h (Tmax)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Tmax
PK parameters for TB511 and Pembrolizumab combination (half-life from 0 to 24 h (t1/2)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination half-life (t1/2)
PK parameters for TB511 and Pembrolizumab combination (Clearance from 0 to 24 h (CL/F)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination CL/F
PK parameters for TB511 and Pembrolizumab combination (Volume of distribution from 0 to 24 h (Vd/F)) [Time Frame: Day 1 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Vd/F
PK parameters for TB511 and Pembrolizumab combination (Area Under the Curve from 0 to 24 h at steady-state (AUCss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUCss
PK parameters for TB511 and Pembrolizumab combination (AUC to the Last Measurable Concentration from 0 to 24 h at steady-state (AUClast ss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUClast, ss
PK parameters for TB511 and Pembrolizumab combination (Area under the plasma concentration-time curve extrapolated to infinity from 0 to 24 h at steady-state (AUCinf, ss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination AUCinf, ss
PK parameters for TB511 and Pembrolizumab combination (Peak Plasma Concentration from 0 to 24 h at steady-state (Cmax ss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Cmax, ss
PK parameters for TB511 and Pembrolizumab combination (Time to Obtain Maximum Plasma Concentration from 0 to 24 h at steady-state (Tmax, ss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Tmax, ss
PK parameters for TB511 and Pembrolizumab combination (half-life from 0 to 24 h at steady-state (t1/2, ss)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination half-life (t1/2, ss)
PK parameters for TB511 and Pembrolizumab combination (Clearance from 0 to 24 h at steady-state (CL, ss/F)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination CL, ss/F
PK parameters for TB511 and Pembrolizumab combination (Volume of distribution from 0 to 24 h at steady-state (Vd, ss/F)) [Time Frame: Day 21 of first 1 cycle] | 2 years
  Determine TB511 and Pembrolizumab combination Vd, ss/F

OTHER OUTCOMES:
Phase I clinical trial-Exploratory Objectives-Biomaker evaluation-class • To compare the changes in biomarker levels of TB511 monotherapy. • To evaluate immunogenicity by measuring anti-drug antibodies against TB511 | 1 year
  Phase I Clinical Trial: 3 to 6 subjects per dose group : Compare changes of the biomarker from the value before TB511 treatment (screening visit) to the post-treatment value (Day 21).
  Tumor tissue-ELISA-CD18, CD163, TGF-ß1, IL-10, VEGF, IFN-γ, Granzyme B Blood-ELISA-TGF-ß1, VEGF, TNF-α, IFN-γ, IL-2 Flow cytometer (Tcell, NK cell)
  -CD45, CD3(CD45+CD3+: T cells), CD4, IFN-γ (Activation), CD25, CD8, Granzyme B(Activation), CD56 (neededCD45+CD3-CD19-CD56: NK), CD19(CD45+CD3-CD19+: B cell)
Phase I clinical trial-Exploratory Objectives-Biomaker evaluation-method • To compare the changes in biomarker levels of TB511 monotherapy. • To evaluate immunogenicity by measuring anti-drug antibodies against TB511 | 1 year
  From the blood collected, the serum will be separated and aliquoted into a tube and kept in a freezer below - 70°C until delivery to the analysis institution. Each tube will be labeled with a subject enrollment number, sampling date, etc; each label will be affixed with tape before storage in a freezer.
  Tumor tissue biomarkers and blood biomarkers will be analyzed using ELISA and a flow cytometer. Tumor tissues will be placed in PBS and crushed using a homogenizer. After centrifuge, the supernatant will be used for ELISA analysis.
  Blood samples will be divided into two: whole blood samples for the flow cytometer and plasma samples for ELISA analysis. Blood and tumor tissues will be analyzed by an external analysis institution. For sample handling and analysis methods, refer to the separately provided manual and the analysis protocol and SOPs of the analysis institution.
Phase I clinical trial-Exploratory Objectives-Anti-drug antibody evaluation • To compare the changes in biomarker levels of TB511 monotherapy. • To evaluate immunogenicity by measuring anti-drug antibodies against TB511 | 1 year
  From the blood collected, the serum will be separated and aliquoted into a tube and kept in a freezer below -70°C until delivery to the analysis institution. Each tube will be labeled with a subject enrollment number, sampling date, etc; each label will be affixed with tape before storage in a freezer.
  ADA to TB511 will be analyzed using ELISA. For ADA analysis, ADA to TB511 will be obtained and sent to an external analysis institution (Bio Infra) together with TB511 capture antibody for analysis. For sample handling and analysis methods for ADA analysis, refer to the separately provided manual and the analysis protocol and SOPs of the analysis institution.
Phase IIa clinical trial-Exploratory Objectives-Biomaker evaluation-class | 2 years
  Biomarker evaluation Phase IIa Clinical Trial: Approximately 20 subjects per cohort (Cohort 1: Approximately 20 subjects, Cohort 2: Approximately 20 subjects) : Compare changes of the biomarker from the value before TB511 treatment (screening visit) to the post-treatment value (Day 21).
  Tumor tissue-ELISA-CD18, CD163, TGF-ß1, IL-10, VEGF, IFN-γ, Granzyme B Blood-ELISA-TGF-ß1, VEGF, TNF-α, IFN-γ, IL-2 Flow cytometer (Tcell, NK cell)
  -CD45, CD3(CD45+CD3+: T cells), CD4, IFN-γ (Activation), CD25, CD8, Granzyme B(Activation), CD56 (CD45+CD3-CD19-CD56: NK), CD19(CD45+CD3-CD19+: B cell)
Phase IIa clinical trial-Exploratory Objectives-Biomaker evaluation-method | 2 years
  From the blood collected, the serum will be separated and aliquoted into a tube and kept in a freezer below - 70°C until delivery to the analysis institution. Each tube will be labeled with a subject enrollment number, sampling date, etc; each label will be affixed with tape before storage in a freezer.
  Tumor tissue biomarkers and blood biomarkers will be analyzed using ELISA and a flow cytometer. Tumor tissues will be placed in PBS and crushed using a homogenizer. After centrifuge, the supernatant will be used for ELISA analysis.
  Blood samples will be divided into two: whole blood samples for the flow cytometer and plasma samples for ELISA analysis. Blood and tumor tissues will be analyzed by an external analysis institution. For sample handling and analysis methods, refer to the separately provided manual and the analysis protocol and SOPs of the analysis institution.
Phase IIa clinical trial-Exploratory Objectives-Anti-drug antibody evaluation | 2 years
  From the blood collected, the serum will be separated and aliquoted into a tube and kept in a freezer below -70°C until delivery to the analysis institution. Each tube will be labeled with a subject enrollment number, sampling date, etc; each label will be affixed with tape before storage in a freezer.
  ADA to TB511 will be analyzed using ELISA. For ADA analysis, ADA to TB511 will be obtained and sent to an external analysis institution (Bio Infra) together with TB511 capture antibody for analysis. For sample handling and analysis methods for ADA analysis, refer to the separately provided manual and the analysis protocol and SOPs of the analysis institution.

IPD SHARING:
Plan to Share IPD: No